CLINICAL TRIAL: NCT06279832
Title: Radiomics and Radiogenomics Models to Predict Molecular Integrated Risk Classes and Prognostic Factors in Endometrial Cancer ID: ROMANTIC STUDY
Brief Title: Radiomics and Radiogenomics Models to Predict Molecular Integrated Risk Classes and Prognostic Factors in Endometrial Cancer.
Acronym: Romantic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Fanfani Francesco, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3994
Record Dates: First submitted 2023-12-15; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Endometrial Cancer
Keywords: Radiomic; Ultrasound; MRI; Molecular sequencing; Radiogenomic; Omic analyses; molecular classification
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: As far as the sample size concerns, the number of images required for the analysis are a figure of at least 100 positive cases (15). We considered as positive patients with a favorable prognostic profile according to PORTEC-4a and also low and intermediate risk class according to ESGO/ESTRO/ESP 2020 recommendations.Therefore, we estimate to enroll at least 1000 patients in order to reach the 100 positive cases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcriptomic analyses (Experimental)
  Interventions: Other: trascriptomic profiling

INTERVENTIONS:
Other: trascriptomic profiling — The mutational and copy number analyses will be complemented by transcriptomic profiling. RNA will be extracted from FFPE samples using miRNAeasy FFPE kit (Qiagen) and checked for quality and quantify by 2100 Bioanalyzer instrument (Agilent) and Qubit Fluorometer (ThermoFisher), respectively. Transcriptome analyses will be performed by RNA-seq. We will apply total RNAseq using the Illumina® TruSeq Stranded Total RNA workflow that provides a solution allowing the detection of whole transcriptome, splicing variants, and transcript fusions of human RNA isolated from FFPE samples. Libraries will be run using the Illumina's Novaseq6000 system, with a least 50 millions of reads/sample, the minimum read depth for the correct evaluation of low expressed transcripts.

SUMMARY:
The aim is to develop radiogenomics models to stratify patients into three main risk categories (Favorable, Intermediate, and Unfavorable) according to the ProMisE model (9) and use these models to predict the most prognostically relevant EC histopathological features (i.e. FIGO stage, degree of tumor differentiation, histotype, LVSI status, myometrial and cervical invasion, lymph node metastases).

These models would support clinicians in personalizing surgical and adjuvant treatment choice among the options considered by the international guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of primary endometrial cancer (endometrioid, clear cell, serous, mixed, any grade)
* FIGO stage IA-IB
* Formalin-fixed, paraffin-embedded (FFPE) tissue at the diagnosis available - Availability of preoperative MRI scans in dicom (.dcm) format
* Availability of preoperative US images in dicom (.dcm) format
* Availability of preoperative CT-scan images in dicom (.dcm) format (optional)
* Available clinical information (e.g. baseline information, surgery, adjuvant therapy, median follow up period 24 months)

Exclusion Criteria:

* Metastatic cancer to the uterus (not primary EC)
* Uterine sarcoma
* Conservative surgery
* FIGO stage > II
* Formalin-fixed, paraffin-embedded (FFPE) tissue at the diagnosis not available
* Patients without available MRI, US or CT-scan images on digital media
* Clinical information not available or incomplete
* Any other malignancy in the previous 5 years or synchronous
* Patients aged under 18 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Predictive value of the model | up to one year
  Receiver operating characteristic (ROC) curve and 95% confidence interval (CI) will be performed to determine cut-off values for the studied quantitative variables.

SECONDARY OUTCOMES:
Validity of the model | up to one year
  To test the validity of different clinical and ultrasound variables Sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) will be determined

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCSS, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: No